CLINICAL TRIAL: NCT02814149
Title: Esthetic, Clinical and Radiographic Outcomes of Immediate Implant Placement and Delayed Implant Placement in the Anterior Region of the Maxilla
Brief Title: Esthetic, Clinical and Radiographic Outcomes of Immediate and Delayed Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Liu, post graduate, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XinL
Record Dates: First submitted 2016-06-15; First posted 2016-06-27 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Jaw, Edentulous, Partially; Acquired Absence of Single Tooth
Keywords: delayed implant; esthetics; immediate implant; bone augmentation
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 1 implant placement (Active Comparator): Implant is placed immediately following tooth extraction in one surgical procedure
  Interventions: Procedure: Type 1 implant placement
- Type 3 implant placement (Active Comparator): Implant is placed in the site which is left to heal for 3 months following tooth extraction
  Interventions: Procedure: Type 3 implant placement

INTERVENTIONS:
Procedure: Type 1 implant placement — Implant is placed immediately following tooth extraction in one surgical procedure
  Other Names: Immediate implant placement
  Arms: Type 1 implant placement
Procedure: Type 3 implant placement — Implant is placed in the site which is left to heal for 3 months following tooth extraction
  Other Names: Delayed implant placement
  Arms: Type 3 implant placement

SUMMARY:
The aim of this prospective cohort study is to compare the esthetic, clinical and patient-centered outcomes following immediate and delayed implant placement protocols.

DETAILED DESCRIPTION:
Patients are divided into two groups: immediate and delayed implant placement. The investigators are asking subjects to take part in a research study of soft tissue and bone healing around dental implants following tooth extraction. The investigators want to compare how the gums and the bone changes shape with healing in two different scenarios.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and able to understand an informed consent
* Adequate oral hygiene to allow for implant therapy consistent with standards of care.
* Missing a single tooth in the maxillary anterior region
* Presence of adjacent natural teeth

Exclusion Criteria:

* Poor oral hygiene
* Severe parafunctional habits, for example, bruxing and clenching
* Presence of clinically active periodontal disease as expressed by probing pocket depths≥4 mm in combination with bleeding on probing.
* Conditions that might lead to a possibly lowered regenerative capacity of the bone, for example, osteoporosis and Paget's disease
* Pregnant or expecting to be pregnant
* History of drug and alcohol abuse
* History of systemic diseases that would contraindicate oral surgical treatment, for example, uncontrolled diabetes (defined as HBA1c level >7%)
* Radiotherapy in the head and neck area,
* On certain medications like bisphosphonates or steroids currently or within the past three months
* Absence of adjacent teeth
* Unwillingness to return for the follow-up examination
* Smokers (more than 20 cigarettes per day). Subjects smoking <20 cigarettes per day were requested to stop smoking before and after surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Pink and white esthetic scores (PES/WES) | Up to 10 years after baseline
  Baseline will be at the time of implant placement.Pink and white esthetic scores (PES/WES) will be recorded at 0.5, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Radiographic bone volume | Up to 10 years after baseline
  Radiographic bone volume be assessed at pre-operation, 0 ,1.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.

SECONDARY OUTCOMES:
Implant survival | Up to 10 years after baseline
  Implant survival will be assessed at 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Probing depth | Up to 10 years after baseline
  Probing depth will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Modified plaque index | Up to 10 years after baseline
  Modified plaque index will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Modified bleeding index | Up to 10 years after baseline
  Modified bleeding index will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Buccal marginal recession | Up to 10 years after baseline
  Buccal marginal recession will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Papilla volume | Up to 10 years after baseline
  Papilla volume will be assessed at 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Width of keratinized gingiva | Up to 10 years after baseline
  Width of keratinized gingiva will be assessed at 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Visual analogue scale (VAS) | Up to 10 years after baseline
  A questionnaire will be recorded at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Oral health impact profile shortened version (OHIP-I) | Up to 10 years after baseline
  A questionnaire will be recorded at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuofan Chen, Study Director — Sun Yat-sen University
Locations (1):
- Guanghua School of Stomatology Hospital of Stomatology, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rieder D, Eggert J, Krafft T, Weber HP, Wichmann MG, Heckmann SM. Impact of placement and restoration timing on single-implant esthetic outcome - a randomized clinical trial. Clin Oral Implants Res. 2016 Feb;27(2):e80-6. doi: 10.1111/clr.12539. Epub 2014 Dec 12. PMID 25496243
- [Background] Huynh-Ba G, Meister DJ, Hoders AB, Mealey BL, Mills MP, Oates TW, Cochran DL, Prihoda TJ, McMahan CA. Esthetic, clinical and patient-centered outcomes of immediately placed implants (Type 1) and early placed implants (Type 2): preliminary 3-month results of an ongoing randomized controlled clinical trial. Clin Oral Implants Res. 2016 Feb;27(2):241-52. doi: 10.1111/clr.12577. Epub 2015 Mar 10. PMID 25758100